CLINICAL TRIAL: NCT01830868
Title: An Open-label, Multi-centre, Multi-national Post-marketing Non-interventional Observational Study of the Use of Zonisamide (ZNS) in the Adjunctive Treatment of Adult Patients With Partial Onset Seizures Treated With One Antiepileptic Drug (AED) as Baseline Medication
Brief Title: A Post-marketing Observational Study Of The Use Of Zonisamide (ZNS) in the Adjunctive Treatment Of Adult Patients With Partial Onset Seizures (Study E2090-E044-410) (ZOOM)
Status: Completed | Type: Observational
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E2090-E044-410
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2023-06-18 (Actual); Status verified 2018-02

CONDITIONS: Partial Onset Seizures
Keywords: ZNS; AED; Partial Onset Seizures; Retention Rate; Seizure Control; Antiepileptic; Secondary generalization; Seizure freedom rates
MeSH Terms: interventions — Zonisamide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Zonisamide tablets
  Interventions: Drug: Zonisamide tablets

INTERVENTIONS:
Drug: Zonisamide tablets — The recommended initial daily dose is 50 mg in two divided doses. After one week the dose may be increased to 100 mg daily and thereafter the dose may be increased at weekly intervals, in increments of up to 100 mg. Doses of 300 mg to 500 mg per day have been shown to be effective, though some patients, especially those not taking CYP3A4 (cytochrome P450)-inducing agents, may respond to lower doses.
  Other Names: ZNS

SUMMARY:
This is a Non-interventional Prospective Study. Centres will enroll adult patients with partial onset seizures for whom the clinician has decided to initiate ZNS as an adjunctive therapy prior to the decision to take part in this study. Patients to be enrolled into the study are not sufficiently controlled with one dug licensed for the use of monotherapy in partial onset seizures. Patients will be seen at baseline and then during normal clinical visits at intervals which are appropriate to the typical practice of the treating clinician. Patients will be assessed at baseline and then at least 3 and 6 months after the baseline.

DETAILED DESCRIPTION:
Open-label, Multi-centre, Multi-national Post-marketing, Non-interventional Observational Study

ELIGIBILITY:
Inclusion Criteria:

* The decision to prescribe ZNS was made by the physician before and independently of his/her decision to include the patient in the study
* Patients treated with one drug licensed for the use as monotherapy in partial onset seizures
* Based on the physician's clinical judgment, the patient seizure activity is not controlled sufficiently with the current monotherapy and it is in the patient's best interest to be prescribed adjunctive ZNS
* Patient was prescribed ZNS no longer than 2 weeks before baseline
* Treatment with ZNS has to be commenced in line with the drug's license and ZNS SmPC (Summary of Product Characteristics)
* Aged 18 years or older
* Capable of understanding the purpose of the study, fully informed and having given written informed consent.

Exclusion Criteria:

* Patients that have started ZNS outside the approved SmPC at enrolment
* Simultaneous participation in an interventional clinical trial and/or taking an investigational drug
* Any form of substance abuse, psychiatric disorder or condition which, in the opinion of the investigator, may complicate communication with the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients With Partial Onset Seizures
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Retention Rate of Zonisamide (ZNS) after 6 months from Baseline | Up to 6 months
  The retention rate or the proportion of patients still receiving ZNS after 6 months will be assessed. At each of the two visits after 3 months and 6 months (final assessment or early discontinuation), the clinician will record whether the patient is still on ZNS treatment, or whether treatment has been discontinued.

SECONDARY OUTCOMES:
Change in Seizure Frequency after 3 and 6 months from Baseline | Baseline, 3 months and 6 months
  Change in overall seizure frequency calculated as absolute and percent changes after 3 and 6 months from baseline compared to the seizure frequency 3 months before introduction of ZNS.

CONTACTS AND LOCATIONS:
Overall Officials: Hajo Hamer, Dr., Principal Investigator — Universitatsklinikum Erlangen, Schwabachanlage 6, 91054 Erlangen, Germany
Locations (37):
- Ried, Austria
- Hillerød, Denmark
- Germany (33):
  - Asperg
  - Baesweiler
  - Berlin
  - Bielefeld
  - Dortmund
  - Eisenach
  - Erbach im Odenwald
  - Erlangen
  - Fürth
  - Gladenbach
  - Hamburg
  - Haßfurt
  - Jülich
  - Kastellaun
  - Lage
  - Lappersdorf
  - Lauf
  - Lohr a. Main
  - Malchin
  - Mönchengladbach
  - München
  - Neuburg an der Donau
  - Neusäß
  - Osnabrück
  - Remscheid
  - Saarbrücken
  - Schorndorf
  - Schwäbisch Gmünd
  - Senftenberg
  - Stralsund
  - Stuttgart
  - Ulm
  - Velen
- Drammen, Norway
- Stockholm, Sweden